CLINICAL TRIAL: NCT01103947
Title: A Comparison of the Efficiency of the New EcoAnaesthesia Facemask With a Standard Facemask During Induction of Anesthesia
Brief Title: EcoAnaesthesia Facemask Versus Standard Facemask During Anesthesia Induction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to finalize funding
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: UoL IRB 09.0588
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia Induction
Keywords: Anesthesia induction; Facemask; surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EcoAnesthesia Mask first (Active Comparator): Both the "standard adult facemask" (Portex Adult, USA) and the new facemask (EcoAnesthesia Mask, Intersurgical, Inc., Liverpool, NY, USA) will be tested in each patient for three minutes. The order of usage of each mask will be randomly assigned to each patient. This group will receive the EcoAnesthesia Mask first.
  Interventions: Device: EcoAnaesthesia facemask first; Device: Portex Adult (Standard) facemask second
- Standard mask first (Active Comparator): Both the "standard adult facemask" (Portex Adult, USA) and the new facemask (EcoAnesthesia Mask, Intersurgical, Inc., Liverpool, NY, USA) will be tested in each patient for three minutes. The order of usage of each mask will be randomly assigned to each patient. Patients in this arm will receive the standard mask first.
  Interventions: Device: Portex Adult (Standard) facemask first; Device: EcoAnesthesia facemask second

INTERVENTIONS:
Device: EcoAnaesthesia facemask first — The trial facemask will be used before the standard one.
  Arms: EcoAnesthesia Mask first
Device: Portex Adult (Standard) facemask first — The standard facemask will be applied before the trial device.
  Arms: Standard mask first
Device: Portex Adult (Standard) facemask second — The standard facemask will be applied after the trial device
  Arms: EcoAnesthesia Mask first
Device: EcoAnesthesia facemask second — The trial facemask will be used after the standard one.
  Arms: Standard mask first

SUMMARY:
This study will evaluate the efficiency of the EcoAnesthesia mask and its advantages over the standard facemask used in our practice. The satisfaction by the anesthesia provider and its ease of use may change the standard practice in airway management. In addition to these additional effects on patient safety, the facemask is affordable and may reduce the environmental burden of anesthesia waste.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class 1-2
* Undergoing elective surgery
* Aged between 18 and 75 years

Exclusion Criteria:

* Severe acute or chronic lung disease requiring oxygen-therapy;
* Hiatus hernia with gastro-esophageal reflux or other esophageal or gastric abnormalities that require a rapid sequence induction;
* Food intake within the last 6 hours or clear fluid intake within 2 hours prior to surgery;
* Ischemic or congenital heart disease;
* Pregnancy (confirmed by a pregnancy test);
* Patient is scheduled for regional anesthesia and denies conductance of general anesthesia during the surgical procedure;
* Known difficult intubation in the past.
* Difficult Mask Ventilation. Patients having any two of the criteria listed below will be Categorized as "Difficult Mask Ventilation (DMV)" (5,13,14) and will be excluded from enrollment. All others will be classified as "Normal." Age > 55 BMI > 26 kg/m2 Lack of teeth Presence of beard History of snoring Limited mandibular protrusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
End-tidal oxygen concentration | three minutes
  End-tidal oxygen concentration after 3 minutes with the mask that the patient was first randomized to use.

SECONDARY OUTCOMES:
Maximum airway pressure | End of 3 minutes with each mask
  Maximum airway pressure, which will be necessary to reach a tidal volume of at least 6 ml/kg every minute during the 3 minutes of mask ventilation with each device.

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Obal, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Background] Kheterpal S, Martin L, Shanks AM, Tremper KK. Prediction and outcomes of impossible mask ventilation: a review of 50,000 anesthetics. Anesthesiology. 2009 Apr;110(4):891-7. doi: 10.1097/ALN.0b013e31819b5b87. PMID 19293691